CLINICAL TRIAL: NCT00195741
Title: Phase III, Randomized, Placebo-Controlled, Double-Blind, Parallel-Group, Multi-Center Study Designed to Evaluate the Safety and Efficacy of Prophylactic Depakote ER in the Treatment of Adolescent Migraine
Brief Title: The Safety and Efficacy of Divalproex Sodium Extended-Release Tablets in Migraine Prophylaxis: A Study in Adolescents
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M02-488
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2007-02-08 (Estimated); Status verified 2007-02

CONDITIONS: Migraine
Keywords: Migraine; Depakote ER
MeSH Terms: conditions — Migraine Disorders | interventions — Valproic Acid

INTERVENTIONS:
Drug: divalproex sodium

SUMMARY:
The purpose of this study is to determine whether Depakote ER is safe and effective in the reduction of occurrence of migraine headaches in adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Subject and subject's legal representative have voluntarily signed and dated an IRB-approved informed assent form and an IRB-approved informed consent form, respectively, before any study-specific procedures or tests are performed, including the discontinuation of any prohibited medications
* Subject is male or a non-pregnant, non-lactating female;
* Subject is between 12 and 17 years of age, inclusive, at randomization;
* Subject weighs between 77 lbs (i.e., 35 kg) and 220 lbs (i.e., 100 kg) inclusive;
* Subject currently has migraine headaches diagnosed according to the International Headache Society (IHS) diagnostic criteria occurring at an average frequency of at least 3, but no more than 12, migraine headaches per month during the 3 months prior to screening. Migraine headaches separated by a headache-free interval of < 48 hours will be considered one migraine headache in assessing this criterion;
* Subject's initial onset of migraine headache precedes the Screening Visit by at least 12 months;
* Subject is judged to be in generally good health based on the results of a medical history, physical examination, 12-lead electrocardiogram (ECG), and laboratory profile. When the Screening and Baseline Visits are combined as described in Section 5.1, continuing participation in the Baseline Phase will be contingent upon laboratory and ECG results. Any repeat laboratory testing must be completed in consultation with the Abbott Medical Monitor prior to randomization.

Experimental Phase

* The following criteria define eligibility for subject enrollment in the

Experimental Phase and subsequent randomization and study drug assignment:

* Subject experienced at least 3, but no more than 12, migraine headaches (separated by headache-free intervals of at least 48 hours), diagnosed according to the IHS diagnostic criteria,6 during the 4-week Baseline Phase of the study; and
* Subject is still eligible for the study based on Baseline Phase inclusion criteria.

Exclusion Criteria Baseline Phase

* History of allergic reaction or significant sensitivity to valproate or similar drugs;
* History of noncompliance with medication or medical instructions;
* Previously randomized in this study;
* Recent (previous 6 months) history of drug and/or alcohol abuse or has a positive urine drug screen, at the Screening Visit, for drugs of abuse (e.g., amphetamines, barbiturates, benzodiazepines, cocaine, opiates, and phencyclidine [PCP]);
* Female, of childbearing potential, and not using an effective method of birth control (e.g., total sexual abstinence or contraceptives);
* History of cluster headaches (see Appendix G, Diagnostic Criteria for Headaches), seizure disorder, or suspected history of seizure disorder;
* History of headaches of any type occurring on 15 or more days per month, on average, or uses medications excessively for headaches (e.g., regularly taking medication on more than 10 days per month);
* Failed more than 2 adequate regimens of prophylactic antimigraine medications, including antiepilepsy drug(s) (e.g., gabapentin, topiramate) or 1 adequate regimen of valproate;
* Use of any prophylactic antimigraine medication within a period equivalent to < 5 half-lives of that medication before entering the Baseline Phase;
* Daily use of any analgesic, ergotamine preparation, or nonsteroidal anti- inflammatory agent (see Appendix J, Examples of Prohibited Medications);
* Use of the following medication classes or any specific drug listed below:

  * anticoagulants
  * antidepressants
  * antiepileptics
  * antipsychotics
  * benzodiazepines
  * beta-adrenergic blocking agents
  * calcium channel antagonists
  * cimetidine
  * corticosteroids
  * cyproheptadine
  * erythromycin
  * ethosuximide
  * lithium salts
  * methysergide
  * phenobarbital
  * pemoline
  * rifampin
  * tolbutamide
  * or zidovudine
* Use of valproate within 30 days prior to screening;
* Use of aspirin and/or any aspirin-containing product (e.g., Excedrin Migraine, Pepto-Bismol, Alka Seltzer) within 5 half-lives prior to randomization or at any time during the Experimental Phase of the study;
* Use of stimulants for Attention-Deficit Hyperactivity Disorder (ADHD) (with the exception of pemoline, Cylert) where a stable treatment regimen has not been established for a minimum of at least 2 months prior to screening or the treatment regimen that has been established is at risk of changing sometime during the trial;
* Any serious medical or psychiatric disorder(s) that may confound the interpretation of the results from this study;
* Central nervous system (CNS) neoplasm, CNS infection, demyelinating disease, degenerative neurological disease, or any progressive CNS disease;
* History of encephalopathy, hepatitis, pancreatitis, or urea-cycle disorder or any underlying condition/disease, which might interfere with study drug absorption or completion of study drug therapy evaluation throughout the duration of the trial;
* Screening laboratory results indicate the presence of Hepatitis B surface antigen (HBSAG), or Hepatitis C antibody or known history of any positive test result for HIV;
* Screening laboratory results indicate: Platelet count </= 100,000/uL ALT or AST >/= 2 times Upper Limit of Normal (ULN);
* Receipt of an investigational drug within 30 days prior to study drug administration or scheduled to receive any other investigational drug anytime during the study; or
* For any reason, subject is considered by the investigator to be an unsuitable candidate to receive Depakote or to participate in this study. Experimental Phase
* Subjects exhibiting any of the following will be ineligible:
* A positive pregnancy test result on Study Day 1;
* Failure to properly maintain the Headache and Medication Diary, during the Baseline phase, to the extent that headache occurrences cannot be determined, due to noncompliance;
* Excessive use of symptomatic medication(s) during the Baseline Phase (e.g., regularly taking medication on more than 10 days per month); or
* Ineligibility for the study based on the Baseline Phase exclusion criteria.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300
Dates: Start 2003-05

PRIMARY OUTCOMES:
Reduction from baseline in 4-week migraine headache rate

SECONDARY OUTCOMES:
Migraine headache rate in last 4 weeks of study
Percent reduction from baseline
Percent of subjects with > 75% reduction in migraine headache rate

CONTACTS AND LOCATIONS:
Overall Officials: Global Medical Information 800-633-9110, Study Director — Abbott
Locations (1):
- Global Medical Information - Abbott, North Chicago, Illinois, United States